CLINICAL TRIAL: NCT03319082
Title: A Phase IV Observational Registry to Assess the Safety and Durability of Effect of Corneal Collagen Cross-linking With Photrexa Viscous, Photrexa, and the KXL System in Patients With Corneal Ectasia Following Refractive Surgery
Brief Title: Observational Registry to Assess the Durability of Effect of CXL in Patients With Corneal Ectasia After Refractive Surgery
Acronym: CXL
Status: Recruiting | Type: Observational
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ACP-KXL-401
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Corneal Ectasia
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CXL Group: Patients with corneal ectasia following refractive surgery who had corneal collagen cross-linking in one or both eyes according to the Photrexa Viscous and Photrexa prescribing information
  Interventions: Combination Product: Corneal Collagen Cross-linking

INTERVENTIONS:
Combination Product: Corneal Collagen Cross-linking — Photrexa Viscous (riboflavin 5'-phosphate in 20% dextran ophthalmic solution), Photrexa (riboflavin 5'-phosphate ophthalmic solution), and the KXL System (UV Irradiation).

SUMMARY:
The objectives of this post market registry are to evaluate the safety and durability of treatment effect up to 3 years following cross-linking performed with Photrexa Viscous (riboflavin 5'- phosphate in 20% dextran ophthalmic solution), Photrexa (riboflavin 5'- phosphate ophthalmic solution), and the KXL System in patients with corneal ectasia following refractive surgery.

DETAILED DESCRIPTION:
Approximately 200 patients who are planning to undergo or have undergone CXL for the treatment of corneal ectasia following refractive surgery in one or both eyes according to the prescribing information in the Photrexa Viscous and Photrexa Package Insert could be enrolled. Patients will be followed for safety and effectiveness at Months 3, 6, 12, 24 and 36 following cross-linking treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age, male or female, of any race;
2. Provide written informed consent and sign a HIPAA form;
3. Willingness and ability to follow all instructions and comply with schedule for study visits;
4. Have a diagnosis of corneal ectasia post-refractive surgery (such as LASIK, PRK);
5. Planning to undergo (or have undergone within the past 90 days) corneal collagen cross-linking with PHOTREXA VISCOUS/ PHOTREXA and the KXL System, per the prescribing information (NOTE: Complete treatment and follow-up data, including any product-related events at time of procedure through the time of enrollment must be available);
6. For females capable of becoming pregnant, agree to have urine pregnancy testing performed prior to enrolling in the registry; must not be pregnant or lactating.

Exclusion Criteria:

1. If female, be pregnant, nursing, or have a positive urine pregnancy test prior to enrollment in the registry;
2. The Investigator may exclude or discontinue any patient for any sound medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with corneal ectasia following refractive surgery who are planning to undergo or have undergone corneal collagen cross-linking in one or both eyes according to the Photrexa Viscous and Photrexa prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Kmax | 36 months
  Change from pretreatment baseline in maximum corneal curvature
BCVA | 36 month
  Change from pretreatment baseline in BCVA

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, Study Director — Glaukos Corporation
Locations (11):
- United States (11):
  - Stanford University School of Medicine, Palo Alto, California
  - Chu Vision Institute, P.A., Bloomington, Minnesota
  - Vance Thompson Vision - MT, Bozeman, Montana
  - Vance Thompson Vision - ND, West Fargo, North Dakota
  - Comprehensive EyeCare of Central Ohio, Westerville, Ohio
  - Vantage Eye Care, LLC, Bala-Cynwyd, Pennsylvania
  - Carolina Cataract & Laser Center, Ladson, South Carolina
  - Slade & Baker Vision, Houston, Texas
  - Hoopes Vision, Draper, Utah
  - See Clearly Vision Group, McLean, Virginia
  - Northwest Eye Surgeons, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hersh PS, Stulting RD, Muller D, Durrie DS, Rajpal RK; U.S. Crosslinking Study Group. U.S. Multicenter Clinical Trial of Corneal Collagen Crosslinking for Treatment of Corneal Ectasia after Refractive Surgery. Ophthalmology. 2017 Oct;124(10):1475-1484. doi: 10.1016/j.ophtha.2017.05.036. Epub 2017 Jun 24. PMID 28655538
- See also: U.S. Multicenter Clinical Trial of Corneal Collagen Crosslinking for Treatment of Corneal Ectasia after Refractive Surgery — https://www.ncbi.nlm.nih.gov/pubmed/?term=peter+hersh